CLINICAL TRIAL: NCT01028989
Title: A Reduced Carbohydrate Diet Intervention for PCOS
Brief Title: A Reduced Carbohydrate Diet Intervention for Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Barbara Gower, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: F090407003; 1R01HD054960-01A2 (NIH)
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Insulin; Diet; Glycemic Load
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reduced Glycemic Load Diet (Other): 36-40% fat; 40-42% carbohydrate; 18-22% protein
  Glycemic Load <=46 per 1000 calories
  Interventions: Dietary Supplement: Reduced Glycemic Load Diet
- Standard Diet (Other): 25-27% fat; 55-57% carbohydrate; 18-22% protein
  Glycemic Load >=77 per 1000 calories
  Interventions: Dietary Supplement: Standard Diet

INTERVENTIONS:
Dietary Supplement: Reduced Glycemic Load Diet — 36-40% fat; 40-42% carbohydrate; 18-22% protein
  Glycemic Load <=46 per 1000 calories
  Arms: Reduced Glycemic Load Diet
Dietary Supplement: Standard Diet — 25-27% fat; 55-57% carbohydrate; 18-22% protein
  Glycemic Load >=77 per 1000 calories
  Arms: Standard Diet

SUMMARY:
Polycystic ovary syndrome (PCOS) affects 5-10% of women of reproductive age, and is associated with infertility, risk for obesity and type 2 diabetes, and impaired quality of life. The elevated insulin characteristic of PCOS is likely to play a major role in its symptoms. Manipulation of dietary carbohydrate quantity and quality (glycemic load; GL) may lower insulin and improve both reproductive and metabolic outcomes. The purpose of this study is to determine if a lower GL diet intervention is more effective than a standard (STD) diet in improving reproductive and metabolic outcomes of women with PCOS in the absence of weight loss.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a heterogeneous syndrome affecting 5-10% of women of reproductive age. It is characterized by elevated circulating insulin, reduced insulin sensitivity, infertility, hyperandrogenism, and a multitude of symptoms that result in a decreased quality of life. The elevated insulin characteristic of PCOS is likely to play a major role in its pathogenesis by reducing insulin sensitivity and stimulating testosterone (T) production and increasing its free fraction. Although many women with PCOS are overweight/obese (10-50%), those who are non-obese suffer from the same symptoms as their obese counterparts. Thus, it is likely that the metabolic disturbances associated with PCOS predispose to weight gain, which in turn exacerbates PCOS by worsening insulin resistance. Manipulation of dietary carbohydrate quantity and quality (glycemic load; GL) may lower insulin and improve both reproductive and metabolic outcomes. No study has tested the efficacy of a lower GL diet among non-obese women with PCOS.

The Specific Aim of this proposal is to determine if a lower GL diet intervention is more effective than a standard (STD) diet in improving reproductive and metabolic outcomes of women with PCOS (both normal-weight and overweight/obese). We hypothesize that, in the absence of weight change, the lower GL diet will be more effective than the STD diet in decreasing insulin secretion, increasing insulin sensitivity, decreasing free T, decreasing fat from metabolically harmful sites, decreasing inflammation, and improving menstrual cyclicity and ovulation. Further, the lower GL diet will increase perceived fullness and decrease hunger, effects mediated via gut hormones.

Development of a diet that optimizes reproductive and metabolic health among women with PCOS will reduce reliance on pharmacologic treatments and improve quality of life, even in the absence of weight loss. This project is novel in being the first to conduct a highly controlled nutrition intervention in non-obese women with PCOS under weight stable conditions, utilizing robust measures of insulin secretion and action, fat distribution, inflammation, hunger/fullness, the gut hormone profile, and reproductive function. The results from this study can be used as a starting point from which to explore optimal diets for overweight women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PCOS
* Body mass index 18.5-35 kg/m2

Exclusion Criteria:

* Cushing's syndrome
* Type 1 or 2 diabetes
* Self-reported claustrophobia
* Androgenic tumors or adrenal hyperplasia
* Hyperprolactinemia
* Implanted metal items
* Use of metformin or other diabetes drug
* Women using oral contraceptives will not be excluded, but will be required to discontinue use of these agents 3 months prior to testing.

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2009-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Improving reproductive and metabolic outcomes of women with PCOS | 8 weeks

SECONDARY OUTCOMES:
The lower Glycemic Load diet will increase perceived fullness and decrease hunger, effects mediated via gut hormones. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A Gower, PhD, Principal Investigator — University of Alabama at Birmingham; Fernando Ovalle, MD, Principal Investigator — University of Alabama at Birmingham; G Wright Bates, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Douglas CC, Gower BA, Darnell BE, Ovalle F, Oster RA, Azziz R. Role of diet in the treatment of polycystic ovary syndrome. Fertil Steril. 2006 Mar;85(3):679-88. doi: 10.1016/j.fertnstert.2005.08.045. PMID 16500338
- [Derived] Hoover SE, Gower BA, Cedillo YE, Chandler-Laney PC, Deemer SE, Goss AM. Changes in Ghrelin and Glucagon following a Low Glycemic Load Diet in Women with PCOS. J Clin Endocrinol Metab. 2021 Apr 23;106(5):e2151-e2161. doi: 10.1210/clinem/dgab028. PMID 33491091
- [Derived] Gower BA, Goss AM. A lower-carbohydrate, higher-fat diet reduces abdominal and intermuscular fat and increases insulin sensitivity in adults at risk of type 2 diabetes. J Nutr. 2015 Jan;145(1):177S-83S. doi: 10.3945/jn.114.195065. Epub 2014 Dec 3. PMID 25527677